CLINICAL TRIAL: NCT05929391
Title: The Effectiveness of Methods for Removing Residual Orthodontic Adhesive From Debonded Metal Attachments: A Randomized Clinical Trial
Brief Title: Effectiveness of Methods to Remove Residual Orthodontic Adhevsie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Saja Saeed Mutar, College of Dentistry/University of Baghdad, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: recycling orthodontic
Record Dates: First submitted 2023-06-08; First posted 2023-07-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Orthodontic Appliance Complication
Keywords: Recycling, Sandblasting, Metal Bracket.

STUDY DESIGN:
Intervention Model Description: split-mouth, cross-quadrant
Who Masked: Participant, Care Provider
Masking Description: The attachments will carry out by main investigator who give each side coded key then the attachments will be rebond by blind specialist. The participants will be blinded to group assignment and interventions (double-blinded trial).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sandblasted group (T1) (Experimental): the side of mouth patient that receives fixed orthodontic appliance that renewed by sandblast
  Interventions: Procedure: Recycling orthodontic brackets
- control group (T3) (Placebo Comparator): the side of mouth patient that receives new fixed orthodontic appliance.
  Interventions: Procedure: Recycling orthodontic brackets
- tungsten bur group (T0) (Experimental): the side of mouth patient that receives fixed orthodontic appliance that renewed by tungsten bur.
  Interventions: Procedure: Recycling orthodontic brackets
- control group (T2) (Placebo Comparator): the side of mouth patient that receives new fixed orthodontic appliance.
  Interventions: Procedure: Recycling orthodontic brackets

INTERVENTIONS:
Procedure: Recycling orthodontic brackets — T0: The adhesive removal will be performed by high-speed hand piece with tungsten carbide bur. the bur will be changed every five attachments. T1: Control group of T0. T2: The adhesive removal will be performed by sandblasting via Micro-etcher.
  T3: Control group of T2.

SUMMARY:
The aim of this study is to compare the clinical efficacy of different residual orthodontic adhesive removing methods for rebonding debonded metal attachments.

DETAILED DESCRIPTION:
1. To evaluate and compare the bond failure rates of rebonded brackets using two methods to remove the adhesive remnant and comparing them with contralateral teeth.
2. To evaluate and compare the bond failure rates of rebonded brackets between different quadrants and arches.
3. To evaluate and compare the bond failure rates of rebonded molar tubes using two methods to remove the adhesive remnant and comparing them with contralateral teeth.
4. To evaluate and compare the bond failure rates of rebonded molar tubes between different quadrants and arches.

ELIGIBILITY:
Inclusion Criteria:

1. Patients need metal fixed orthodontic appliance treatment;
2. Complete set of permanent dentition with fully erupted teeth on both arches;
3. Intact teeth and mainly their buccal surfaces are free from caries, fillings, or gingival hyperplasia;
4. No occlusal interferences that can affect the ideal position of attachments, especially in the lower arch.

Exclusion Criteria:

1. patients have crown, missing teeth, or craniofacial anomalies.
2. patients have congenital enamel defects specially their buccal surface.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The number of bonding failures will be compared using the chi-square test. | baselines
  evaluate and compare the bond failure rates. different quadrants and arches.To evaluate and compare the bond failure rates of rebonded attachments(brackets and molar tubes)using two methods (Tungsten carbide bur and sandblasting)) to remove the adhesive remnant and comparing them with contralateral teeth.

SECONDARY OUTCOMES:
The bonding failure between each quadrant will be compared by one way ANOVA. | bsaelines
  evaluate and compare the bond failure rates. different quadrants and arches.

CONTACTS AND LOCATIONS:
Locations (1):
- 2 private dental clinics in Iraq and special center in Karbala., Baghdad, Iraq

REFERENCES:
- [Background] Ahmed T, Rahman NA, Alam MK. Assessment of in vivo bond strength studies of the orthodontic bracket-adhesive system: A systematic review. Eur J Dent. 2018 Oct-Dec;12(4):602-609. doi: 10.4103/ejd.ejd_22_18. PMID 30369810
- [Background] Alessandri Bonetti G, Zanarini M, Incerti Parenti S, Lattuca M, Marchionni S, Gatto MR. Evaluation of enamel surfaces after bracket debonding: an in-vivo study with scanning electron microscopy. Am J Orthod Dentofacial Orthop. 2011 Nov;140(5):696-702. doi: 10.1016/j.ajodo.2011.02.027. PMID 22051490
- [Background] Eminkahyagil N, Arman A, Cetinsahin A, Karabulut E. Effect of resin-removal methods on enamel and shear bond strength of rebonded brackets. Angle Orthod. 2006 Mar;76(2):314-21. doi: 10.1043/0003-3219(2006)076[0314:EORMOE]2.0.CO;2. PMID 16539561